CLINICAL TRIAL: NCT04485598
Title: Genetic Identification of Monogenic Disorders in Early-onset Stroke Using Targeted Next Generation Sequencing Panel
Acronym: MDEOS
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Executive Vice-President, Beijing Tiantan Hospital
Other Study IDs: CNSR3-ngs-eos
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Stroke, Acute; Transient Ischemic Attack; Single-gene Disorders
Keywords: Stroke; Transient Ischemic Attack; Targeted sequencing panel; Early-onset
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Genomic DNA was extracted from peripheral blood leukocytes,
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study was designed as a multicenter multiracial prospective observational study of acute ischemic stroke and TIA patients across china. The purpose of this study is to determine the monogenic disorders incidence of Chinese early-onset stroke patients. We plan to consecutively enroll more than 500 patients with early-onset stroke(in the 18- to 45-year age range) admitted in stroke units within 7 days after symptoms onset in participating centers. These early-onset stroke patients are referred for targeted sequencing using 'cerebrovascular disease panel'. By analyzing the sequencing results, we intend to identify monogenic causes causing early-onset stroke and develop clinical algorithms that might assist the clinician in deciding in which early-onset stroke patients testing for monogenic causes of stroke.

DETAILED DESCRIPTION:
The study was designed as a multicenter multiracial prospective observational study of acute ischemic stroke and TIA patients across china. The purpose of this study is to determine the monogenic disorders incidence of Chinese early-onset stroke patients. We plan to consecutively enroll more than 500 patients with early-onset stroke(in the 18- to 45-year age range) admitted in stroke units within 7 days after symptoms onset in participating centers. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be referred for targeted sequencing using 'cerebrovascular disease panel'. When one or multiple pathogenic or possible pathogenic exonic mutations are found, a Sanger Sequencing (SS) on somatic DNA from peripheral blood leukocyte of the index case and affected relatives will be performed for the screening of the same mutations. And the sporadic patient's mutations will be checked by SS in the unaffected family members. By analyzing the sequencing results, we intend to identify monogenic causes causing early-onset stroke and develop clinical algorithms that might assist the clinician in deciding in which early-onset stroke patients testing for monogenic causes of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Female or male aged ≥ 18 years and ≤ 45 years.
* Acute ischemic stroke or Transient ischemic attack((Neurological deficit attributed to focal brain ischemia, with resolution of the deficit within 24 hours of symptom onset) patients that can be enrolled within 7 days of symptoms onset defined by the"last see normal"principle.

Exclusion Criteria:

* Asymptomatic brain infarction
* Neurological deficit due to causes other than ischemic stroke or TIA

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Acute ischemic stroke or Transient ischemic attack patients from participating centers over China that can be enrolled within 7 days of symptoms onset defined by the"last see normal"principle.Female or male aged ≥ 18 years and ≤ 45 years.
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2015-08-21 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with certain etiologic diagnosis established with targeted sequencing | day 0
  Percentage of patients with certain etiologic diagnosis established with targeted sequencing

SECONDARY OUTCOMES:
Obtained read depth according to number of pooled samples | day 0
  Obtained read depth according to number of pooled samples
Percentage of patients with variant with unknown significance | day 0
  Percentage of patients with variant with unknown significance, needing supplementary analyses to prove its involvement in early-onset stroke
Clinical phenotype for each gene for which a causal mutation is identified by targeted sequencing panel | day 0
  Clinical phenotype for each gene for which a causal mutation is identified by targeted sequencing panel
Time of analysis of NGS raw data | 30 days
  Time of analysis of NGS raw data
Incidence of certain single-gene disorders in early-onset stroke patients | day 0
  Incidence of certain single-gene disorders in early-onset stroke patients

CONTACTS AND LOCATIONS:
Overall Officials: Wei Li, M.D, Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality, China